CLINICAL TRIAL: NCT00258661
Title: Multicenter Osteopathic Pneumonia Study in the Elderly (MOPSE)
Brief Title: Is Osteopathic Manipulative Treatment (OMT) Beneficial for Elderly Patients Hospitalized With Pneumonia?
Acronym: MOPSE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: A.T. Still University of Health Sciences (Other)
Collaborators: Brentwood Foundation (Other); Colorado Springs Osteopathic Foundation (Other); Foundation for Osteopathic Health Services (Maryland) (Unknown); Muskegon General Osteopathic Foundation (Michigan) (Unknown); Northwest Oklahoma Osteopathic Foundation (Oklahoma) (Unknown); Osteopathic Founders Foundation (Oklahoma) (Unknown); Osteopathic Institute of the South (Georgia) (Unknown); Osteopathic Heritage Foundations (Other); Quad City Osteopathic Foundation (Iowa) (Unknown)
Responsible Party: Brian F Degenhardt, DO, A.T. Still University - A.T. Still Research Institute
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Treatment
Other Study IDs: 501-202
Record Dates: First submitted 2005-11-23; First posted 2005-11-28 (Estimated); Last update posted 2018-10-04 (Actual); Status verified 2018-10

CONDITIONS: Pneumonia
Keywords: Pneumonia; Osteopathic; Manipulation; Multi-center; Elderly
MeSH Terms: conditions — Pneumonia | interventions — Manipulation, Osteopathic

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Osteopathic Manipulative Treatment (Experimental): 10-minute standardized OMT protocol + 5-minute nonstandardized component, twice daily for duration of hospitalization
  Interventions: Procedure: Osteopathic Manipulative Treatment
- Light-touch Treatment (Sham Comparator): 10-minute standardized light-touch protocol (designed to mimic OMT standardized protocol) + 5-minute auscultation of carotid bruits, heart, and lungs, twice daily for duration of hospitalization
  Interventions: Procedure: Light-touch Treatment
- Conventional Care Only (No Intervention): No intervention specific to the research study provided. Only conventional treatment as per attending physician orders.

INTERVENTIONS:
Procedure: Osteopathic Manipulative Treatment — In addition to conventional treatment for pneumonia, a 10-minute standardized OMT protocol + 5-minute nonstandardized component was performed twice daily for the duration of hospitalization.
  Other Names: OMT; OMM; Osteopathic Manipulative Medicine; Manipulation
  Arms: Osteopathic Manipulative Treatment
Procedure: Light-touch Treatment — In addition to conventional treatment for pneumonia, a 10-minute standardized light-touch protocol (designed to mimic OMT standardized protocol) + 5-minute auscultation of carotid bruits, heart, and lungs was performed twice daily for the duration of hospitalization.
  Other Names: Sham manipulation; Placebo manipulation
  Arms: Light-touch Treatment

SUMMARY:
Osteopathic Manipulative Treatment (OMT) were used in the 1800s and 1900s to treat pneumonia before the introduction of antibiotics in the mid-1900s. The purpose of this study is to determine if OMT, when used in conjunction with antibiotics and other usual care, will improve the recovery of elderly pneumonia patients.

DETAILED DESCRIPTION:
This study is a multi-center study conducted across five sites in the United States to determine the efficacy of combining Osteopathic Manipulative Treatment(OMT)with antibiotics as a treatment regimen for elderly patients with pneumonia. The study is a prospective, randomized, controlled clinical trial, in which 360 subjects will be randomly assigned to three different groups to test the primary hypothesis that the combination of OMT and antibiotics will decrease the length of hospital stay for elderly patients with pneumonia. The first group (OMT Group) will receive a series of eight osteopathic manipulative techniques in combination with conventional antibiotic care. The second group (Light Touch Control Group) will receive a light touch mimic treatment in combination with conventional antibiotic care to control for the doctor-patient interaction. The third group (Conventional Care Only Group) will receive only the conventional antibiotic care normally given to elderly patients with pneumonia. The first two groups will receive two 15-20 minute treatments per day, at least six hours apart, for the duration of their stay in the acute care facility.

The primary outcomes for measuring efficacy are: Length of Hospital Stay, Time to Clinical Stability, and Rate of Symptomatic and Functional Recovery. The secondary outcomes are: duration of IV and oral antibiotic usage in the hospital, number of complications and deaths secondary to pneumonia, re-admission rate within 60 days of hospitalization admission date, duration and severity of fever, duration and severity of leukocytosis, and patient satisfaction.

ELIGIBILITY:
Inclusion Criteria:

* 50 Years old or older
* Subject is hospitalized in an acute care facility
* Subject must exhibit at least two of the classic symptoms of pneumonia, to include:
* Respiration Rate greater than or equal to 25 respirations per minute
* New or increased cough
* Fever greater than or equal to 100.4 degrees F (38 degrees C)
* Pleuritic chest pain
* Worsening of mental or functional status
* Leukocytosis (WBC greater than 12,000 cells per cubic millimeter)
* New or increased physical findings (rales, wheezing, bronchial breath sounds)

Exclusion Criteria:

* Lung abscess
* Advancing pulmonary fibrosis
* Bronchiectasis
* Pulmonary tuberculosis
* Lung Cancer
* Metastatic malignancy
* Uncontrolled metabolic bone disease that places subject at risk for pathologic bone fracture (i.e. Paget's Disease or hypoparathyroidism)
* Acute or unhealed rib or vertebral fracture
* History of pathologic bone fracture
* Previous participants as subject in the study
* Respiratory failure (intubation)

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 406 (Actual)
Dates: Start 2004-03; Primary Completion 2007-04 (Actual); Study Completion 2007-04 (Actual)

PRIMARY OUTCOMES:
Length of Hospital Stay | End of hospital stay
  Number of days from admission order to discharge order
Time to Clinical Stability | Daily for the duration of the hospital stay
  Halm EA, Fine MJ, Marrie TJ, Coley CM, Kapoor WN, Obrosky DS, et al.:
  Time to clinical stability in patients hospitalized with community-acquired pneumonia: implications for practice guidelines. JAMA 1998, 279:1452-1457
Symptomatic and Functional Recovery Score | 14, 30, and 60 days post-admission
  Metlay JP, Fine MJ, Schulz R, Marrie TJ, Coley CM, Kapoor WN, et al.:
  Measuring symptomatic and functional recovery in patients with communityacquired pneumonia. J Gen Intern Med 1997, 12:423-430

SECONDARY OUTCOMES:
Duration of IV and oral antibiotic usage in the hospital
Number of complications and deaths secondary to pneumonia
Duration and severity of fever
Duration and severity of leukocytosis
Patient Satisfaction

CONTACTS AND LOCATIONS:
Overall Officials: Donald R Noll, D.O., FACOI, Principal Investigator — A.T. Still University
Locations (7):
- United States (7):
  - Mount Clemens General Hospital, Mount Clemens, Michigan
  - Northeast Regional Medical Center, Kirksville, Missouri
  - UNDNJ in association with Kennedy Memorial Hospitals- University Medical Center, Stratford, New Jersey
  - Doctors Hospital, Columbus, Ohio
  - John Peter Smith Health Network, Fort Worth, Texas
  - Plaza Medical Center, Fort Worth, Texas
  - UNTHSC Osteopathic Medical Center, Fort Worth, Texas

REFERENCES:
- [Background] Noll DR, Degenhardt BF, Fossum C, Hensel K. Clinical and research protocol for osteopathic manipulative treatment of elderly patients with pneumonia. J Am Osteopath Assoc. 2008 Sep;108(9):508-16. PMID 18806080
- [Result] Noll DR, Degenhardt BF, Morley TF, Blais FX, Hortos KA, Hensel K, Johnson JC, Pasta DJ, Stoll ST. Efficacy of osteopathic manipulation as an adjunctive treatment for hospitalized patients with pneumonia: a randomized controlled trial. Osteopath Med Prim Care. 2010 Mar 19;4:2. doi: 10.1186/1750-4732-4-2. PMID 20302619
- [Derived] Noll DR, Degenhardt BF, Johnson JC. Multicenter Osteopathic Pneumonia Study in the Elderly: Subgroup Analysis on Hospital Length of Stay, Ventilator-Dependent Respiratory Failure Rate, and In-hospital Mortality Rate. J Am Osteopath Assoc. 2016 Sep 1;116(9):574-87. doi: 10.7556/jaoa.2016.117. PMID 27571294